CLINICAL TRIAL: NCT05063019
Title: Adding Value of Magnetic Resonance Imaging and Magnetic Resonance Enterography for the Pre-operative Assessment of Imaging Peritoneal Cancer Index in Patients With Peritoneal Carcinomatosis
Brief Title: Role of Magnetic Resonance Enterography for Predicting Peritoneal Cancer Index
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202100965A3
Record Dates: First submitted 2021-09-13; First posted 2021-09-30 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-09

CONDITIONS: Hyperthermic Intraperitoneal Chemotherapy; Cytoreductive Surgery; Peritoneal Carcinomatosis
Keywords: Hyperthermic Intraperitoneal Chemotherapy; Cytoreductive Surgery; Peritoneal Cancer Index; Magnetic Resonance Enterography
MeSH Terms: conditions — Peritoneal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnetic resonance imaging and enterography following computed tomography (Experimental): Magnetic resonance imaging and enterography will be performed after computed tomography but before surgery.
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Magnetic resonance imaging and enterography before surgery

SUMMARY:
This is a prospective observational study which will recruit 90 participants over a three-year period to investigate whether adding magnetic resonance imaging and enterography to routine computed tomography study can better predict the extend of peritoneal carcinomatosis over computed tomography alone.

DETAILED DESCRIPTION:
Hyperthermic Intraperitoneal Chemotherapy (HIPEC) is a new option for patients with peritoneal carcinomatosis and the effectiveness of HIPEC depends on the extend of disease. Currently, pre-operative imaging peritoneal cancer index (PCI) is used to predict the intraoperative tumor extend and completeness of cytoreduction. However, the investigators' previous study and literature review show that imaging PCI usually underestimated intraoperative PCI, resulting in subsequent Open-Close operation. The investigators hypothesize that magnetic resonance imaging (MRI) is a better predictor of the intra-operative PCI than computed tomography (CT), and MR Enterography can better represent tumor deposits in the small intestine. This study aims to test whether the addition of MRI and MR Enterography to CT study improves the prediction performance of the intraoperative PCI and completeness of optimal cytoreduction over CT alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with peritoneal carcinomatosis diagnosed by computed tomography
* Schedule for operation at our institute

Exclusion Criteria:

* Age < 20 years old
* Renal function impairment or acute renal failure
* Contraindications for magnetic resonance imaging
* Primary tumor not origins from colorectal cancer, gastric cancer or ovarian cancer

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Predicting intraoperative PCI scores for patients with peritoneal carcinomatosis, using MR Enterography and CT | 36 months
  The Sugarbaker's Peritoneal Cancer Index scores according to the MR enterography and CT images will be calculated pre-operatively and will be compared to the standard PCI scores obtained during operation. Basically, the scoring system divides the abdominopelvic cavity into 13 separate regions, and each region is scored 0-3 points as follows: 0 point, the absence of tumor; 1 point, tumors < 0.5 cm in diameter; 2 points, tumors 0.5-5 cm in diameter; 3 points, tumors > 5 cm in diameter.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ni Lin, MA, Principal Investigator — Chang Gung Memorial Hospital, Chiayi, Taiwan
Locations (1):
- Chang Gung Memorial Hospital, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers.